CLINICAL TRIAL: NCT00465244
Title: Seizure Therapy With Intravenous Levetiracetam and Lorazepam
Acronym: STILL
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inability to recruit subjects
Sponsor: Massachusetts General Hospital (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Joshua N. Goldstein, MD, PhD, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STILL
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Seizures
Keywords: Prehospital and ED seizures
MeSH Terms: conditions — Seizures | interventions — Levetiracetam; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Levetiracetam 1 g IV + Lorazepam 2 mg IV
  Interventions: Drug: Levetiracetam 1 g IV + Lorazepam 2 mg IV
- 2 (Other): Placebo + Lorazepam 3 mg IV
  Interventions: Drug: Placebo + Lorazepam 3 mg IV

INTERVENTIONS:
Drug: Levetiracetam 1 g IV + Lorazepam 2 mg IV — Levetiracetam 1 g IV + Lorazepam 2 mg IV
  Arms: 1
Drug: Placebo + Lorazepam 3 mg IV — Placebo + Lorazepam 3 mg IV
  Arms: 2

SUMMARY:
The overarching aim of STILL is assessment of IV LEV in the management of seizures in the ED setting. The main study endpoints are considered in the two patient groups of interest (SE and non-SE):

* For non-SE patients, STILL will compare IV LEV vs. the current standard-care of placebo, with respect to the following questions:
* Does IV LEV administration result in lower seizure duration and/or recurrence rate than does administration of placebo? (Ho: No difference in seizure duration or recurrence rates between the two groups.)
* Is IV LEV associated with a different rate of significant side effects than placebo? (Ho: No difference in significant side effect rates between the two groups.)
* For SE patients, STILL will compare [IV LEV + lorazepam 2mg] vs. [lorazepam 3 mg], with respect to the following questions:
* Does addition of IV LEV to a BZD allow for a BZD-sparing effect (i.e. achievement of seizure control with lower dose of BZD)? (Ho: No difference in seizure duration and/or recurrence rates between the two groups.)
* Is IV LEV + lower-dose BZD associated with a different rate of significant side effects than the higher-dose BZD administered as monotherapy? (Ho: No difference in significant side effect rates between the two groups.)

DETAILED DESCRIPTION:
The study will enroll adults (age at least 18 years) in the EDs of MGH or BWH. Patients will be classified, depending upon their clinical presentation, into the SE group or the non-SE group. The total enrollment projected for non-SE patients is 150; the total enrollment projected for SE patients is 200. It is expected that at least 3 years may be required to enroll the requisite number of patients.

Patients are eligible for study enrollment if they have had a seizure, and if they do not have known pregnancy or renal failure, and if they are not known to be breastfeeding. Hypotension is the only other exclusion criteria for the study. There are no other contraindications to study enrollment.

Patients evaluated at the MGH/BWH EDs for seizures may arrive by private vehicle or ambulance. A "STILL" pager will be activated by ED physicians upon notification of impending ambulance arrival with a suspected seizure patient (SE or non-SE); the pager can also be activated after patient arrival at the ED by ambulance or private vehicle.

Upon patient arrival to the ED, standard stabilization will be provided. If the patient is determined to have had a seizure, or if the patient is currently seizing, an IV will be placed (if not already present) in line with standard ED care. For the patient to be eligible for STILL, the seizure must have occurred within an hour of ED arrival.

Care providers will make a determination as to whether patients are eligible, using a checklist readily available in the ED. For patients who are determined to be eligible, the care providers will indicate whether patients are in the "SE" or "non-SE" arm - the study groups are hereafter denoted SE and non-SE.

STILL medications will be stored in the ED with other medications, so that they are readily available to care providers. The STILL medications will be in a separate section of the automated drug dispenser units in the ED. STILL medications will be subdivided as to whether patients are in the SE or non-SE arms. In each of the two subsections (SE and non-SE) of the EDs' automated drug dispensers will be one box of study medications. Thus, the ED will always have on hand, sufficient study medications to enroll one patient in either the SE or non-SE arm. The randomization procedures to determine the contents of the study medication boxes will be done in the Research Pharmacy, so no randomization needs to occur prior to treatment in the ED. The study boxes will have unique identifier numbers, which will then be reported back to the Research Pharmacy after the study medications have been administered; the Research Pharmacy thus will have track of which study patients received which study boxes (and which medication regimens). This approach to patient allocation and drug dispensing and tracking is consistent with current mechanisms for enrolling patients in Partners IRB-approved studies in the MGH/BWH EDs.

Inside the SE partition in the ED box will be a syringe containing lorazepam (concentration: 2 mg/mL) in either a 2 mg or 3 mg dose; an extra volume of inactive diluent will be added to the 2 mg dose so that the volume (1.5 mL) is that same in each syringe. In a manner consistent with previous/ongoing Partners IRB-approved studies in the ED, the syringe will be labeled "lorazepam - 2mg or 3mg." Also in the SE compartment of the drug dispenser will be an infusion set labeled "levetiracetam 1.5g or placebo." Thus, for SE patients, care providers will administer two agents from the medication dispenser; patients will receive either [lorazepam 2mg + levetiracetam 1.5 g] or [lorazepam 3mg + placebo]. Care providers will be instructed (by information included with the study drugs) to administer the lorazepam over 1.5-2 minutes (this is in line with standard recommendations that lorazepam be administered at a rate not to exceed 2 mg/min).28, 38 The infusion (i.e. levetiracetam or placebo) will be administered over 5 minutes.

Inside the non-SE partition in the ED box will be an infusion set labeled "levetiracetam 1.5g or placebo." Thus, for non-SE patients, care providers will administer one agent from the medication dispenser; patients will receive either levetiracetam 1.5 g or placebo. Care providers will be instructed (by information included with the study drugs) to administer the infusion over 5 minutes.

The contents of the partitions in the ED drug dispenser will be determined in advance, by a randomization scheme that prevents the need for care providers to make a phone call or otherwise spend time (which they do not have) randomizing patients. When the EDs use study drug from either arm of STILL, they will contact the Research Pharmacy which will replace the used materials and note the patient's medical record number along with the true identity of the study agent(s) administered.

Any adjunctive medication may be administered at the discretion of the treating physicians.

Study endpoints for SE and non-SE patients are outlined in the Detailed Protocol. Briefly, SE analysis will focus on whether seizure recurrence is reduced, and whether respiratory depression and other post-medication vital signs changes occur less frequently in patients receiving LEV and the smaller dose of lorazepam, as compared to those receiving the higher-dose lorazepam alone. For non-SE patients, endpoints will include seizure recurrence as well as quality of the examination and occurrence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* seizure

Exclusion Criteria:

* pregnancy
* renal failure
* hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Seizures | hours
Mental status | hours
Respiratory depression | hours
seizure recurrence | hours

CONTACTS AND LOCATIONS:
Overall Officials: Joshua N. Goldstein, MD, PhD, Principal Investigator — Massachusetts General Hospital